CLINICAL TRIAL: NCT02648919
Title: Phase II Clinical Study of Noni Extract in Men With Very Low Risk or Low Risk Prostate Cancer
Brief Title: Clinical Study of Noni Extract in Men With Very Low Risk or Low Risk Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: University of Hawaii (Other)
Collaborators: University of Hawaii Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUANG-2015-1
Record Dates: First submitted 2015-12-30; First posted 2016-01-07 (Estimated); Results first posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Noni 6,000 mg/day (Experimental): Noni extract 6,000 mg/day (4 capsules with breakfast, 4 capsules with lunch and 4 capsules with dinner)
  Interventions: Drug: Noni extract

INTERVENTIONS:
Drug: Noni extract — Intervention will be administered on an outpatient basis.Six bottles containing 60 capsules will be dispensed to all participants upon enrollment. Then 12 bottles (at 30-day visit) and 18 bottles (at 3, 6 and 9 month visits) will be dispensed to all participants.
  Other Names: Healing Noni

SUMMARY:
The purpose of this study is to evaluate the effects of Noni extract in men diagnosed with very low risk or low risk prostate cancer

DETAILED DESCRIPTION:
Efficacy and safety of Noni extract will be assessed in an estimated sample size of 30 subjects. Efficacy will be measured by the induction of favorable gene expression changes on Oncotype Dx Prostate Cancer Test after 12 months of intervention with Noni extract (6,000 mg/day). Other efficacy endpoints include the incidence of tumor progression after 12 months of intervention with Noni extract and serum PSA doubling time. Safety measurements will include the incidence and severity of adverse events, effects on angiogenesis (CD34), cell proliferation (Ki-67), and apoptosis (TUNEL) in prostate tissue biopsy samples from Month 12

ELIGIBILITY:
Inclusion Criteria:

1. Men with a diagnosis of very low risk (<5% risk of disease relapse after primary treatment, criteria; cT1c, Gleason <6, PSA < 10 ng/mL, fewer than 3 positive biopsy cores < 50% cancer in any core, PSA density < 0.15 ng/mL/g); low risk (10% risk of disease relapse after primary treatment, criteria; cT1-2a, Gleason <6, PSA < 10 ng/mL) prostate cancer
2. Very low risk and low risk groups will be confirmed by Oncotype DX prostate cancer test and provided a Genomic Prostate Score (GPS)
3. 55 years of age and older (>/= 55 years) at the time of informed consent
4. No evidence of extraprostatic disease on 3T multiparametric pelvic MRI
5. No baseline PT/PTT abnormalities, coagulopathies, or who are on any blood thinners.
6. ECOG performance status 0-2
7. Participants must have normal organ and marrow function as demonstrated by the following parameters being:

   * complete blood count (CBC) - no clinically significant findings
   * complete metabolic profile (CMP) - no clinically significant findings
8. Willing to comply with proposed visit and treatment schedule
9. Able to understand and willing to sign a written informed consent document

Exclusion Criteria:

1. Prior history of treated prostate cancer
2. Concomitant use of medications that are known CYP3A4 substrates
3. Use of medications or supplements that are known to affect PSA within 30 days prior to informed consent, including toremifene citrate, finasteride, testosterone, dehydroepiandrosterone (DHEA) or other testosterone-like supplements. No dutasteride within 90 days prior to informed consent
4. Consumption of any concomitant nutritional, herbal supplements, and antioxidants should be taken under the discretion of the investigator. The following foods/supplements are prohibited at least 7 days prior to initiation of and during study treatment:

   * St. John's wort or hyperforin (potent CYP3A4 enzyme inducer)
   * Grapefruit juice (potent cytochrome P450 CYP3A4 enzyme inhibitor)
5. Use of any blood thinners.
6. Consumption or use of any Noni or Noni-containing products
7. History of renal or hepatic disease, including history of hepatitis B or C. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or any psychological, familial, sociological or other concomitant condition that would not allow adequate compliance with the study protocol
8. Participation in any other investigational study or use of any other investigational agents within 30 days prior to study entry
9. History of allergic reactions attributed to Noni or other compounds of similar chemical or biologic composition to Noni, or the inactive components present in Noni capsules.

Min Age: 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Huang, PharmD, Principal Investigator — Faculty
Locations (1):
- University of Hawaii Cancer Center, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Issell BF, Franke A, Fielding RM. Pharmacokinetic study of Noni fruit extract. J Diet Suppl. 2008;5(4):373-82. doi: 10.1080/19390210802519671. PMID 22436097

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Noni 6,000 mg/Day
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Noni 6,000 mg/Day: Noni extract 6,000 mg/day (4 capsules with breakfast, 4 capsules with lunch and 4 capsules with dinner)
  Noni extract: Intervention will be administered on an outpatient basis. Six bottles containing 60 capsules will be dispensed to all participants upon enrollment. Then 12 bottles (at 30-day visit) and 18 bottles (at 3, 6 and 9 month visits) will be dispensed to all participants.
Arm/Group | Noni 6,000 mg/Day
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 68 [59 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Compare Genomic Prostate Score (GPS) in Prostatic Tumors
Description: Exploring gene expression changes on Oncotype DX Genomic Prostate Score (GPS). The Oncotype DX assay is a clinically validated 17-gene genomic assay that provides a genomic prostate score (GPS; scale 0-100) measuring the heterogeneous nature of prostate tumors. A higher score means a higher risk of disease. Unfortunately, Genomic Health was unable to run the assay on 12-month prostate biopsy samples in which active cancer was not identified therefore we only have baseline data.
Time Frame: Change from screening and at 12 months or early termination
Measure: Number; unit: scores on a scale
Arm/Group | Noni 6,000 mg/Day
Number analyzed (Participants) | 6
scores on a scale
  GPS Pt 1 Baseline | 37
  GPS Pt 2 Baseline | 34
  GPS Pt 3 Baseline | 17
  GPS Pt 4 Baseline | 36
  GPS Pt 5 Baseline | 38
  GPS Pt 6 Baseline | 39

2. Primary Outcome: Number of Positive Cores Associated With Participants Disease Progression of Prostate Cancer
Description: Measure tumor size at screening and compare after 12 months of study participation. Disease progression will be identified by either an increase in Gleason score, increase in positive cores, and/or an increase in tumor volume.
Time Frame: Change from screening and at 12 months or early termination
Measure: Number; unit: positive cores
Arm/Group | Noni 6,000 mg/Day
Number analyzed (Participants) | 6
positive cores
  Positive Cores pre therapy Pt 1 | 1
  Positive Core post therapy Pt 1 | 6
  Positive Cores pre therapy Pt 2 | 2
  Positive Cores post therapy Pt 2 | 5
  Positive Cores pre therapy Pt 3 | 1
  Positive Cores post therapy Pt 3 | 3
  Positive Cores pre therapy Pt 4 | 1
  Positive Cores post therapy Pt 4 | 0
  Positive Cores pre therapy Pt 5 | 1
  Positive Cores post therapy Pt 5 | 0
  Positive Cores pre therapy Pt 6 | 1
  Positive Cores post therapy Pt 6 | 0

3. Secondary Outcome: Effects of Noni Extract on Serum Prostate Specific Antigen (PSA) Levels
Description: Comparing the serum Prostate Specific Antigen (PSA) test levels for the duration of the trial in men diagnosed with very low risk or low risk prostate cancer. Measure the duration of time it takes for a subjects Prostate specific antigen level to double.
Time Frame: Baseline and 9 months
Measure: Number; unit: ng/mL
Arm/Group | Noni 6,000 mg/Day
Number analyzed (Participants) | 6
ng/mL
  PSA Baseline Pt 1 | 4.4
  PSA Baseline Pt 2 | 5.4
  PSA Baseline Pt 3 | 7.3
  PSA Baseline Pt 4 | 9.7
  PSA Baseline Pt 5 | 6.9
  PSA Baseline Pt 6 | 7.9
  PSA 9 Month Pt 1 | 5.7
  PSA 9 Month Pt 2 | 9.6
  PSA 9 Month Pt 3 | 10.2
  PSA 9 Month Pt 4 | 6.9
  PSA 9 Month Pt 5 | 8.1
  PSA 9 Month Pt 6 | 7.7

4. Secondary Outcome: Frequency of Adverse Events
Description: Tolerability of Noni extract in men diagnosed with very low risk or low risk prostate cancer as assessed by CTCAE v4.0
Time Frame: Enrollment, 1, 3, 6, 9, and 12 months, and 7 days post treatment
Measure: Number; unit: Adverse Events Reported
Arm/Group | Noni 6,000 mg/Day
Number analyzed (Participants) | 6
Adverse Events Reported | 3

5. Secondary Outcome: Explore the Molecular Pathways Contributing to the Activities Associated With Noni Extract in the Prostate Cancer (e.g. Cell Proliferation, and Apoptosis in Prostate Tissue Biopsy Samples) Via Immunohistochemistry (IHC) Staining.
Description: Utilizing prostate tissue biopsy samples and serum blood plasma from participants prior to receiving noni extract and after the subject completes 12 months of receiving noni extract. Apoptosis was quantified based on caspase-3 immunostaining. Proliferation was quantified based on Ki-67 immunostaining.
Time Frame: Enrollment and 12 months or at early termination
Measure: Mean (Standard Deviation); unit: percentage of positive cells
Arm/Group | Noni 6,000 mg/Day
Number analyzed (Participants) | 6
percentage of positive cells
  Apoptosis Pre Treatment | 12.2 (3.2)
  Proliferation Pre Treatment | 1.2 (0.3)
  Apoptosis Post Treatment | 10.9 (2.1)
  Proliferation Post Treatment | 1.4 (0.4)

6. Secondary Outcome: Explore the Molecular Pathways Contributing to the Activities Associated With Noni Extract in the Prostate Cancer (e.g., Angiogenesis) in Prostate Tissue Biopsy Samples) Via Immunohistochemistry (IHC) Staining.
Description: Utilizing prostate tissue biopsy samples and serum blood plasma from participants prior to receiving noni extract and after the subject completes 12 months of receiving noni extract. MVD, a surrogate for angiogenesis, was quantified based on CD-31 immunostaining.
Time Frame: Enrollment and 12 months or at early termination
Measure: Mean (Standard Deviation); unit: microvessel/mm^2
Arm/Group | Noni 6,000 mg/Day
Number analyzed (Participants) | 6
microvessel/mm^2
  MVD Pre Treatment | 60.5 (18.1)
  MVD Post Treatment | 41.2 (9.5)

ADVERSE EVENTS:
Time Frame: The incidence and severity of adverse events occurring during the study intervention will be reported. The period of time the subject will be receiving study intervention is 12 months. Participants will have study visits at Months 1, 3, 6, 9, and 12 months and at each time point will be assessed for adverse events. All reported Adverse events were followed until resolution.
Groups:
- Noni 6,000 mg/Day: Noni extract 6,000 mg/day (4 capsules, 3 times per day)
  Noni extract: Intervention will be administered on an outpatient basis.Six bottles containing 60 capsules will be dispensed to all participants upon enrollment. Then 12 bottles (at 30-day visit) and 18 bottles (at 3, 6 and 9 month visits) will be dispensed to all participants.
Arm/Group | Noni 6,000 mg/Day
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Noni 6,000 mg/Day (N=6)
diarrhea (Gastrointestinal disorders) | 1 (2) — Subject experienced grade 3 diarrhea after 1 month of study intervention introduction. This same subject had recurrence of grade 3 diarrhea 5 months after the initial event reported.
depression (Psychiatric disorders) | 1 (1) — subject with history of depression was admitted to hospital for 1 week due to depression with psychotic features

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-02-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT02648919/Prot_SAP_000.pdf
  • Informed Consent Form (2017-02-24): https://cdn.clinicaltrials.gov/large-docs/19/NCT02648919/ICF_001.pdf